CLINICAL TRIAL: NCT03345888
Title: To Compare Predictive Power of End-tidal Carbon Dioxide Between Different Time Line During Resuscitation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20171110PUMCHER
Record Dates: First submitted 2017-11-14; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Resuscitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- resuscitation time line group: The ETCO2 will be arrange in resuscitation time line.
  Interventions: Other: predictive power of end-tidal carbon dioxide
- ETCO2 time line group: The ETCO2 will be arrange in time line which the beginning time is the time of starting to show stable ETCO2 wave.
  Interventions: Other: predictive power of end-tidal carbon dioxide

INTERVENTIONS:
Other: predictive power of end-tidal carbon dioxide — end-tidal carbon dioxide predicts resuscitation outcomes

SUMMARY:
To analyze a multi-center observational study database. to select adult non-traumatic in-hospital cardiac arrest. Review and recored end-tidal carbon dioxide in per minute. Arrange them in different time line. one is in resuscitation time. The other is the time line which the beginning time is the time of starting appearing stable end-tidal carbon dioxide wave.To compare predictive power of end-tidal carbon dioxide between different time line during resuscitation.

ELIGIBILITY:
Inclusion Criteria:

adult non-traumatic in-hospital cardiac arrest patients Exclusion Criteria:1) surrogate decision of Do-Not-Resuscitate (DNR) during CPR; 2) out-of-hospital cardiac arrest (OHCA) patient; 3) trauma as the main reason for medical treatment; 4) child or adolescent patients; 5) Petco2 value was not recorded effectively; 6) delay from initial CPR to starting to record Petco2 exceeded 30 min; and 7) screening by qualified experts. More than three experienced physicians thought that the patient's Petco2 value was too extreme to agree with his/her medical history, and the value was seen as an error and was excluded

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: CPR patient being treated in the emergency department
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2017-11-10 (Actual); Primary Completion 2017-11-15 (Estimated); Study Completion 2017-11-17 (Estimated)

PRIMARY OUTCOMES:
predictive power of ETCO2 is week at the beginning of resuscitation | 1 week
  the later predictive power of ETCO2 is better during 30min resuscitation

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided